CLINICAL TRIAL: NCT01112605
Title: Standard Deviation of the Distance Between the Sural Nerve and Achilles Tendon by Ultrasound
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Omer Mei-Dan, Meir Medical Center
Other Study IDs: MMC09155-09CTIL
Record Dates: First submitted 2010-02-16; First posted 2010-04-28 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: achilles tendon; sural nerve; distance; US; ultrasound; Distance between Sural nerve and the Achilles tendon

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- otherwise healthy persons: healthy persons, no major trauma or surgery of ankle or calves, no bone or muscle disease, age 18-60

SUMMARY:
The purpose of this study is to define the standardization of the distance between the Sural nerve & Achilles tendon, in otherwise healthy persons and athletes.

DETAILED DESCRIPTION:
The distance between the two anatomic structures is measured by US and data is analyzed to define the standardized distance in the population in order to avoid damage to the sural nerve while repairing an Achilles tendon rupture using the percutaneous methode.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 18-60

Exclusion Criteria:

* known bone or muscle disease
* major trauma to the leg or ankle in present or past
* surgery of leg or ankle in the past
* mental disabilities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: otherwise healthy persones, age 18-60, community sample.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
distance between the Sural nerve & the Achilles tendon | day 1
  one time measurment of the distance between the sural nerve & the Achilles tendon, using an US device.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei-Dan, Dr., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel